CLINICAL TRIAL: NCT00449631
Title: Multidrug Resistance After Trabeculectomy With Mitomycin C
Status: Completed | Type: Observational
Sponsor: University of Cologne (Other)
Other Study IDs: Multidrug Resistance
Record Dates: First submitted 2007-03-19; First posted 2007-03-20 (Estimated); Last update posted 2007-03-26 (Estimated); Status verified 2007-03

CONDITIONS: Glaucoma; Trabeculectomy
Keywords: Glaucoma; Drug Resistance, Multiple; Trabeculectomy
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
We investigate whether mitomycin C treatment during previous filtration surgery induces P-glycoprotein expression.

DETAILED DESCRIPTION:
Despite the adjuvant use of mitomycin C during trabeculectomy, short-term and long-term failures still occur. We investigate whether mitomycin C treatment during previous trabeculectomy induces P-glycoprotein expression. Expression of P-glycoprotein is analysed in surgically removed Tenon tissue using immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* patients with planned trabeculectomy for elevated eye pressure
* one third of patients without previous trabeculectomy
* two thirds of patients with previous trabeculectomy (one third with and one third without the use of mitomycin C)

Exclusion Criteria:

* patients not requiring surgery
* patients with planned surgery for elevated eye pressure other than trabeculectomy

Ages: 8 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Arno Hueber, MD, Principal Investigator — University of Cologne
Locations (1):
- The University Hospital of Cologne, Cologne, Germany

REFERENCES:
- [Derived] Hueber A, Esser JM, Kociok N, Welsandt G, Luke C, Roters S, Esser PJ. Mitomycin C induces multidrug resistance in glaucoma surgery. Graefes Arch Clin Exp Ophthalmol. 2008 Feb;246(2):297-304. doi: 10.1007/s00417-007-0695-1. Epub 2007 Oct 13. PMID 17934748